CLINICAL TRIAL: NCT01510821
Title: A Prospective Trial to Investigate Endothelial Dysfunction in Saphenous Vein Grafts Subjected to the Maquet Vasoshield Pressure Limiting Syringe Versus Non-Regulated Vessel Dilation in Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: Investigation of Endothelium in Saphenous Vein Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Maquet Cardiovascular (Industry)
Responsible Party: Principal Investigator, Vinod Thourani, Associate Professor of Surgery, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00049331
Record Dates: First submitted 2011-11-02; First posted 2012-01-18 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Endothelial Function of Saphenous Vein Grafts
Keywords: endoscopic vein harvest; saphenous vein graft; endothelial function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maquet Vasoshield Arm (Experimental): Pressure limiting syringe
  Interventions: Other: Use of Maquet Vasoshield Pressure-limiting syringe on SVG
- Non-regulated Arm (Active Comparator): standard non-regulated syringe
  Interventions: Other: Use of non-regulated syringe on SVG

INTERVENTIONS:
Other: Use of Maquet Vasoshield Pressure-limiting syringe on SVG — Use of Maquet Vasoshield Pressure-limiting syringe on SVG
  Other Names: Maquet device
  Arms: Maquet Vasoshield Arm
Other: Use of non-regulated syringe on SVG — Use of non-regulated syringe on SVG
  Other Names: standard syringe
  Arms: Non-regulated Arm

SUMMARY:
This is a single center prospective study of 30 patients undergoing elective heart bypass surgery (CABG) with at least two vein grafts from the leg (SVG). The purpose of this ex vivo study is to evaluate the function of vein grafts from small tissue samples treated with a pressure syringe and a non-pressure syringe. Syringes are routinely used to flush out the veins in preparation of bypass grafting. It is unknown if different levels of pressure in the syringe affect the vein or damage the vein. Small sections of tissue samples which are normally discarded will be obtained immediately after retrieval from the leg and before grafting to the heart. Tissue samples will be taken to the laboratory for study. There are no clinical endpoints in this study, however, clinical information will be obtained from the Society of Thoracic Surgeons database and will include demographics, risk factors, and perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective coronary artery bypass graft surgery requiring at least 2 saphenous vein grafts

Exclusion Criteria:

* patients undergoing any concomitant surgical procedures

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
SVG vascular contractility | Day of surgery

SECONDARY OUTCOMES:
Nitric oxide metabolite levels | Day of surgery
Major adverse cardiac events | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Thourani, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Cardiothoracic Surgery Research Laboratory, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia